CLINICAL TRIAL: NCT06540157
Title: Investigating the Effectiveness of Binaural Beat Music Combined With Rhythmic Photic Stimulation on Depression, Quality of Life, and Heart Rate Variability in Elderly Patients With Depression
Brief Title: Binaural Beat Music Combined With Rhythmic Photic Stimulation on Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Yang Shang-Yu, Associate professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Asia0725
Record Dates: First submitted 2024-07-25; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBM and RPS group (Experimental): All participants received 20-minute interventions daily from Monday to Friday for 12 weeks.
  Interventions: Other: Binaural Beat Music (BBM) Combined with Rhythmic Photic Stimulation (RPS)
- Sham group (Sham Comparator): All participants received 20-minute interventions daily from Monday to Friday for 12 weeks.
  Interventions: Other: Sham group

INTERVENTIONS:
Other: Binaural Beat Music (BBM) Combined with Rhythmic Photic Stimulation (RPS) — Participants rested on a chair for 10 minutes before the intervention. Participants wore over-ear stereo headphones and RPS glasses, receiving 20 minutes of 10Hz BBM (embedded with classic old songs as mask music) and RPS. The BBM and RPS glasses were purchased from George Szeless's mindLightz.
  Arms: BBM and RPS group
Other: Sham group — Participants rested on a chair for 10 minutes before the intervention. Participants wore the same headphones and RPS glasses as the BBM and RPS group but listened to classic Taiwanese old songs without the 10Hz light stimulation from the RPS glasses.
  Arms: Sham group

SUMMARY:
Background: Previous studies have suggested that non-pharmacological treatments, such as binaural beat music (BBM) and rhythmic photic stimulation (RPS), may help improve depressive symptoms and enhance quality of life. However, their effectiveness in elderly patients with depression remains unclear.

Objectives: This study aims to investigate the effects of combining BBM and RPS on improving depression, quality of life, and heart rate variability (HRV) in elderly patients with depression.

Methods: This study was conducted as a single-blind randomized controlled trial. Forty-eight elderly patients with depression were recruited from a long-term care institution in Taiwan and randomly assigned to either the BBM and RPS group or the Sham group. Participants received 20 minutes of intervention daily, Monday to Friday, for 12 consecutive weeks. During the intervention, participants in the BBM and RPS group listened to 10Hz BBM (embedded with classic old songs) and wore RPS glasses that provided 10Hz light stimulation. In contrast, participants in the Sham group listened to classic old songs and wore RPS glasses without the 10Hz light stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this study were:

A) Diagnosed with major depressive disorder by a psychiatrist and stable for more than six months; B) Aged 65 and above; C) No cognitive impairment, with a Mini-Mental State Examination (MMSE) score above 24 and able to understand the questionnaire content; D) No severe physical illnesses and no significant hearing impairments; E) Not using antidepressants within three months before and during the intervention.

Exclusion Criteria:

* Exclusion criteria included:

A) History of mixed psychiatric disorders, including schizophrenia, bipolar disorder, and dementia; B) Experiencing acute illness (or pain) and unstable physiological conditions; C) History of epilepsy or potential for seizures; D) Substance abuse; E) Participation in electroconvulsive therapy or transcranial electrical stimulation within one month before and during the intervention.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | On Day 84 of the intervention, the researchers conducted the posttest (second test) at the participants' long-term care institution and the test content was the same as the first test. It took about 10 minutes.
  There were 21 questions in the BDI, and a self-rated method was used for participants to fill in their thoughts in the last 2 weeks. A 4-point Likert scale was used. The score range of each question was 0-3 points. A total score of 0-12 points was normal, 14-19 points was mild depression, 20-28 points was moderate depression, and 29-63 points was severe depression.
World Health Organization Quality of Life-BREF (WHOQOL-BREF) | On Day 84 of the intervention, the researchers conducted the posttest (second test) at the participants' long-term care institution and the test content was the same as the first test. It took about 10 minutes.
  The Taiwanese version of WHOQOL-BREF measured quality of life, containing 28 items scored on a 5-point Likert scale. It covered four domains: Physical Health (7 items), Psychological Health (6 items), Social Relationships (4 items), and Environment (9 items). Scores ranged from 4 to 20 points, with higher scores indicating better quality of life.
HRV analyzer | On Day 84 of the intervention, the researchers conducted the posttest (second test) at the participants' long-term care institution and the test content was the same as the first test. It took about 10 minutes.
  HRV (Heart Rate Variability) Measurements:
  Mean heart rate (bpm): This measures the average number of heartbeats per minute.
  SDNN (ms): Standard deviation of all RR intervals, representing the physiological health of the autonomic nervous system. A higher SDNN indicates better physiological health.
  nLF (Normalized Low Frequency, ms²): Reflects sympathetic nervous activity. A higher value indicates greater activity.
  nHF (Normalized High Frequency, ms²): Reflects parasympathetic nervous activity. A higher value indicates greater activity.
  LF/HF (ratio): A marker reflecting the balance between sympathetic and parasympathetic nervous activity.

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Yu Yang, PhD, Study Chair — Asia University
Locations (1):
- Asia Univeraity, Taichung, WuFeng, Taiwan